CLINICAL TRIAL: NCT05912894
Title: Anatomical Variation in Rouvière's Sulcus: a Cross-sectional Study
Brief Title: Anatomical Variation in Rouvière's Sulcus
Status: Not yet recruiting | Type: Observational
Sponsor: University Of Perugia (Other)
Collaborators: Giovanni Domenico Tebala (Unknown); Luca Properzi (Unknown); Nereo Vettoretto (Unknown); Matteo Matteucci (Unknown); Antonio Pesce (Unknown); Carlo Boselli (Unknown); Antonia Rizzuto (Unknown); Augusto Lauro (Unknown)
Responsible Party: Principal Investigator, Roberto Cirocchi, Associate Professor in General Surgery, University Of Perugia
Other Study IDs: AVRS1
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Rouvière's Sulcus
Keywords: Prevalence Rouvière's Sulcus; Anatomical variations Rouvière's Sulcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Videolaparoscopic cholecystectomy: Patients undergoing Videolaparoscopic cholecystectomy
  Interventions: Procedure: Videolaparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Videolaparoscopic cholecystectomy — Evaluation of Rouvière's Sulcus Anatomical Variation.

SUMMARY:
Rouvière's sulcus is a 2-5 cm fissure lying on the lower face of the liver, between the right lobe and caudate process. Due to its extrabiliary location, Rouvière's Sulcus could be used as an anatomical landmark for safe laparoscopic cholecystectomy. In literature there's an high variability about Rouvière Sulcus prevalence and its anatomical variants.

DETAILED DESCRIPTION:
The goal of this observational study is to evaluate the presence of Rouvière Sulcus in patients underwent laparoscopic cholecystectomy. The main questions it aims to answer are the prevalence and the anatomical variations of Rouvière's Sulcus and the variants of Rouvière's Sulcus which are catheghorized according to Singh and Prasad criteria.

The following were considered secondary outcome: operative time expressed in minutes, biliary tract injuries according to Stewart's classification and Vascular injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing videolaparoscopic cholecystectomy

Exclusion Criteria:

* If the lower face of the right hepatic lobe and the main elements of the biliary tract cannot be clearly analyzed patients will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Rouvière's Sulcus | 2 years
Anatomical variations in Rouvière's Sulcus | 2 years
  The variants of the Rouvière's Sulcus are catheghorized by the classification of Singh e Prasad.

SECONDARY OUTCOMES:
Operative time | 2 years
  Time expressed in minutes
Biliary tract injuries | 2 years
  Biliary tract injuries according to Stewart's classification.
Vascular injuries | 2 years
  Vascular injuries.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh M, Prasad N. The anatomy of Rouviere's sulcus as seen during laparoscopic cholecystectomy: A proposed classification. J Minim Access Surg. 2017 Apr-Jun;13(2):89-95. doi: 10.4103/0972-9941.201731. PMID 28281470
- [Background] Stewart L. Iatrogenic biliary injuries: identification, classification, and management. Surg Clin North Am. 2014 Apr;94(2):297-310. doi: 10.1016/j.suc.2014.01.008. PMID 24679422
- [Background] Pesce A, Fabbri N, Feo CV. Vascular injury during laparoscopic cholecystectomy: An often-overlooked complication. World J Gastrointest Surg. 2023 Mar 27;15(3):338-345. doi: 10.4240/wjgs.v15.i3.338. PMID 37032796